CLINICAL TRIAL: NCT01527474
Title: An Open-label Study of Escitalopram in the Treatment of Postpartum Depression
Brief Title: Escitalopram in the Treatment of Postpartum Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BC Women's Hospital & Health Centre (Other)
Responsible Party: Principal Investigator, Dr. Shaila Misri, Principal Investigator, BC Women's Hospital & Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SM1562007
Record Dates: First submitted 2012-02-03; First posted 2012-02-07 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Postpartum Depression
Keywords: postpartum; postpartum depression; PPD; escitalopram
MeSH Terms: conditions — Depression, Postpartum | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: escitalopram — participants will be initiated at a dose of 10mg/day which will be adjusted by the study clinician based on the presences of depressive symptoms and side effects up to a maximum of 20mg/day.

SUMMARY:
This will be an 8-week, open-label trial evaluating the efficacy of escitalopram as monotherapy in the treatment of patients with postpartum depression (PPD). The acute phase of the study will consist of an 8 week treatment phase. Treatment of eligible participants will be initiated at a dose of 10mg/day which will be adjusted by the study clinician based on the presence of depressive symptoms and side effects up to a maximum of 20mg/day.

Study objectives are:

1. to investigate the efficacy of escitalopram in the treatment of PPD.
2. to assess the effects of escitalopram on patients quality of life.

DETAILED DESCRIPTION:
Major Depression Postpartum Onset (PPD) is a chronic relapsing illness which affects not only maternal mood but also the baby and family. Therefore, it is critical to aim for timely intervention once the diagnosis is made. Studies have shown that antidepressant medications are effective in treatment for moderate to severe PPD. Common reasons for noncompliance and discontinuation of antidepressant medications in the postpartum period are the side effects associated with different antidepressants. To choose an antidepressant medication with proven efficacy and a tolerable side effect profile is key in order to maximize adherence to pharmacotherapy.

A number of studies have been published that highlight the efficacy of escitalopram in the treatment of Major Depressive Disorder (MDD). However, there has been no research to date investigating the effectiveness of escitalopram in the treatment of PPD.

Based upon the preliminary clinical observations in our tertiary care program (Provincial Reproductive Mental Health Program) where a postpartum depressed population is frequently treated with antidepressant medications, compliance with escitalopram has been impressive. Therefore, we propose to conduct an open-label study with escitalopram in postpartum depressed, non-lactating mothers to confirm our clinical observation.

Hypotheses:

i) Escitalopram will be effective in the treatment of Postpartum Depression and ii) Escitalopram will be effective in increasing the quality of life of participants.

ELIGIBILITY:
Inclusion Criteria:

* female between the ages of 19 to 40 years of age
* given birth in the last 6 months
* not currently breastfeeding
* meet criteria for Major Depressive Disorder as per the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV TR)
* Montgomery-Asberg Depression Rating Scale (MADRS) score greater than or equal to 25 at enrolment
* able to read and write English
* sign written informed consent to participate in the study.

Exclusion Criteria:

* have a significant risk of suicide according to the investigator's opinion or presents a score of 5 or greater on item 10 (suicidal thoughts) of of the MADRS
* meets DSM-IV-TR criteria for past or current manic or hypomanic episode, past or current psychotic symptoms or disorder, and/or has a history of drug or alcohol abuse/dependence within the last 6 months
* uses the following disallowed recent or concomitant medication within the specified time periods - any antidepressant or any drug used for augmentation of antidepressant action within the last 2 weeks (5 weeks for fluoxetine) prior to baseline, any benzodiazepines or other anxiolytics within the last week prior to baseline, any non-benzodiazepine hypnotics within the last week prior to baseline, oral antipsychotics within 2 weeks or depot antipsychotics within 6 months prior to baseline, serotonergic medicinal products (for example triptans, tryptophan, tramadol) within the last week prior to baseline, psychoactive herbal remedies (for example St. Johns Wort, kava kava, valerian, gingko biloba) within the last 2 weeks prior to baseline, any other drug with potential psychotropic effects within the last 2 weeks prior to baseline, any anticonvulsant drug within the last 2 weeks prior to baseline, or any investigational product within 3 months prior to baseline
* is currently receiving formal cognitive or behavioural therapy, systematic psychotherapy, or plans to initiate such therapy during the study
* current depressive symptoms of the patient are considered by the investigator to have been resistant to two well-conducted antidepressant treatments of at least 6 weeks duration
* has a serious illness or serious sequelae thereof, including liver or renal insufficiency, or a cardiovascular, pulmonary, gastrointestinal, endocrine, neurological (including epilepsy), infectious, neoplastic, or metabolic disturbance (if there is a history of such disease but the condition has been stable for at least one year and is judged by the investigator not to render inclusion unsafe and not to interfere with the patient's participation in the study, the patient may be included.)

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The primary efficacy assessment will be total score on the Montgomery-Asberg Depression Rating Scale (MADRS). | The primary endpoint will be the change from baseline on MADRS total score after 8-weeks of treatment.

SECONDARY OUTCOMES:
The Secondary efficacy assessment will be total score on the short form of the Quality of Life Enjoyment and Satisfaction Questionnaire. | The secondary endpoint will be change from baseline on the Quality of Life Enjoyment and Satisfaction Questionnaire total score after 8-weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Shaila Misri, MD, Principal Investigator — University of British Columbia
Locations (1):
- Reproductive Mental Health Program, BC Women's Hospital, Vancouver, British Columbia, Canada